CLINICAL TRIAL: NCT01368458
Title: A Randomized, Rater-Blind, Controlled, Clinical Trial of Conversion to Antipsychotic Monotherapy vs. Continued Polypharmacy for Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Conversion to Antipsychotic Monotherapy
Acronym: MOPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Joshua Kantrowitz MD, Nathan Kline Institute for Psychiatric Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07I/C31
Record Dates: First submitted 2008-07-01; First posted 2011-06-08 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conversion to mono therapy (Experimental): Conversion from 2 to 1 antipsychotic
  Interventions: Other: Conversion to Antipsychotic Monotherapy
- control (No Intervention): No change in antipsychotics

INTERVENTIONS:
Other: Conversion to Antipsychotic Monotherapy — Patients assigned to the antipsychotic monotherapy group will have the dosage of their secondary (i.e. one due to be reduced) antipsychotic reduced by decreased by approximately 1/3 every 3 weeks. Dosage of the primary antipsychotic will be left unchanged.
  Arms: Conversion to mono therapy

SUMMARY:
This is a 12-week, with a 32-week follow-up, rater-blind, randomized controlled trial to determine whether patients with chronic schizophrenia or schizoaffective disorder receiving two different antipsychotics simultaneously will have any significant change in psychopathology following conversion to antipsychotic monotherapy. Additionally, the effects of conversion to antipsychotic monotherapy will be assessed by neurocognitive tests.

The study will be conducted at the Clinical Research and Evaluation Facility (CREF), a specialized research unit jointly operated by the Nathan S Kline Institute for Psychiatric Research (NKI) and Rockland Psychiatric Center (RPC). Patients will be recruited from the regular in-patient units of RPC and transferred to the CREF. Following baseline assessments, patients will be randomized to continued antipsychotic polypharmacy treatment or to systematic conversion to monotherapy.

Conversion to antipsychotic monotherapy will be assessed across multiple domains of psychopathology using the Positive and Negative Symptom Scale (PANSS). The primary outcome measure is PANSS total score. The secondary outcome measure is time on medication (all-cause dropouts). Mixed Model Repeated Measures (MMRM) will test the hypothesis that conversion to antipsychotic monotherapy will show minimal change from the control group.

DETAILED DESCRIPTION:
Background:

Often, treatment resistant schizophrenia patients are treated with high doses of, or polypharmacy with, antipsychotics, or both. There is a lack of systematic evidence for either practice, and this is not recommended by most treatment guidelines. Often polypharmacy results in dosages well above the recommended upper limit of dosage. Recent studies of antipsychotic utilization, have reported that approximately 10-60% of patients are prescribed at least two antipsychotics.

Moreover, antipsychotic treatment carries substantial risks, including the potential development of tardive dyskinesia or metabolic syndrome. Higher doses may expose patients to more adverse events or consequences without any additional therapeutic benefit. Clear benefits of long-term treatment with antipsychotic polypharmacy have rarely been reported, and there is a void of long term double blind, placebo controlled trials.

Antipsychotic polypharmacy remains common, including patients receiving atypical antipsychotics. To our knowledge, no one has published a study of a systematic, randomized controlled conversion to antipsychotic monotherapy for patients with chronic schizophrenia or schizoaffective disorder receiving atypical antipsychotic polypharmacy.

Design:

Hospitalized patients with DSM-IV-TR schizophrenia or schizoaffective disorder meeting the following criteria: (1) at least two antipsychotics, (2) stable dosages for at least one month prior to baseline, (3) baseline dosages of at least one of the antipsychotics are at least olanzapine 15 mg, ziprasidone 120 mg, quetiapine 500 mg, risperidone 4 mg, aripiprazole 10 mg, paliperidone 6 mg, any dose of clozapine, or any first generation antipsychotic >300 chlorpromazine equivalents.

After a baseline assessment, patients will be randomized to conversion to antipsychotic monotherapy of one of their two antipsychotics or continued on their combination antipsychotic treatment. Other psychotropics will be left unchanged from baseline, and the prescription of a new psychotropic will not be permitted, excepting lorazepam and benztropine as detailed below.

If a patient is randomized to conversion to monotherapy, then the decision of which of the two baseline antipsychotics to continue will occur as follows:

1. If one is clozapine, then clozapine will be continued.
2. In all other cases:

   1. If only one of the antipsychotics is at a dose greater than the above noted doses, then that is one that will be continued.
   2. If both doses are greater than the above noted doses, then there will be a flip of a coin to determine which to continue, with heads equal the one with the higher alphabetic letter and tails equal to the lower.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-64 with a SCID DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder, confirmed by SCID, who are able to give written informed consent and on stable dosages of two antipsychotics for at least one month prior to baseline.

Exclusion Criteria:

* Lack of capacity to give informed consent (capacity is determined by a licensed member of the treatment team)
* unstable medical illness
* use of long acting injectable preparations of antipsychotic medication in the previous two months
* documented failure of previous dose reduction
* current treatment with clozapine
* addition of any new psychotropic in the previous month
* patients who are severely assaultive and in clinical need of more than one antipsychotic for their safe management

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-12; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) total score | 12 weeks
Relapse Rate | 12 weeks

SECONDARY OUTCOMES:
Nurses Observation Scale for Inpatient Evaluation (NOSIE) | 12 weeks
Abnormal Involuntary Movement Scale (AIMS) | 12 weeks
Simpson-Angus Scale (SAS) | 12 weeks
Barnes Akathisia Scale | 12 weeks
MATRICS | 12 weeks
Clinical Global Impression (CGI) | 12 weeks
Weight | 12 weeks
Calgary Depression Scale for Schizophrenia (CDSS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Kantrowitz, MD, Principal Investigator — Nathan Kline Institute